CLINICAL TRIAL: NCT01981473
Title: Anti-tnf Inhibitor Antibody-mediated Blockade Of Drug Efficacy In Rheumatoid Arthritis (Antibody-ra)
Brief Title: Drug Concentration, Immunogenicity, and Efficacy Study in Patients With Rheumatoid Arthritis Currently Treated With Etanercept, Adalimumab, or Infliximab
Acronym: ANTIBODY-RA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801364; ANTIBODY-RA (Other: Alias Study Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; etanercept; adalimumab; infliximab; anti-drug antibody; immunogenicity; drug concentration
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab; Infliximab

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- etanercept: Participants currently receiving etanercept treatment in a clinical setting for a minimum of 6 months and maximum of 24 months prior to study assessment visit.
  Interventions: Other: no intervention
- adalimumab: Participants currently receiving adalimumab treatment in a clinical setting for a minimum of 6 months and maximum of 24 months prior to study assessment visit.
  Interventions: Other: no intervention
- infliximab: Participants currently receiving infliximab treatment in a clinical setting for a minimum of 6 months and maximum of 24 months prior to study assessment visit.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention
  Other Names: Enbrel
  Groups: etanercept
Other: no intervention
  Other Names: Humira
  Groups: adalimumab
Other: no intervention
  Other Names: Remicade
  Groups: infliximab

SUMMARY:
The purpose of this study is to examine the relationship between anti-drug antibodies, serum drug concentrations, and clinical response for rheumatoid arthritis patients being treated with etanercept, adalimumab or infliximab.

DETAILED DESCRIPTION:
cross-sectional Population will be selected through convenience sampling. Patients sequentially visiting the rheumatology clinic for routine care who are receiving etanercept, adalimumab, or infliximab for between 6 and 24 months will be evaluated for eligibility and interest in participation. A maximum of 200 patients per treatment will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of RA based on the 1987 American College of Rheumatology revised criteria
3. Current continuous treatment with either etanercept, adalimumab, or infliximab for a minimum of 6 months and maximum of 24 months.

Exclusion Criteria:

1. Treatment with biosimilar or investigational etanercept, adalimumab, or infliximab within past 6 months.
2. Treatment with any other investigational drugs within past 3 months or five half lives of the drug, whichever is longer.
3. Any medical condition that would interfere with rheumatoid arthritis evaluation or other study assessments (eg, fibromyalgia, lupus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from patients seen in a rheumatology clinical setting who currently treated with etanercept, adalimumab or infliximab for rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (34):
  - Arizona Arthritis & Rheumatology, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology, Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, Sun City, Arizona
  - Mercy Clinic Hot Springs Communities, Hot Springs, Arkansas
  - Sutter Institute for Medical Research, Sacramento, California
  - Arthritis Care Center, Incorporated, San Jose, California
  - Rheumatology Consultants of Delaware dba Delaware Arthritis, Lewes, Delaware
  - Omega Research Consultants, LLC, DeBary, Florida
  - Center for Rheumatology, Immunology, and Arthritis, Fort Lauderdale, Florida
  - Florida Medical Research, Gainesville, Florida
  - Arthritis and Rheumatic Care Center, South Miami, Florida
  - Health Point Medical Group, Inc., Tampa, Florida
  - Northeast Georgia Diagnostic Clinic, LLC, Gainesville, Georgia
  - Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Rheumatology Associates of Baltimore, Baltimore, Maryland
  - Phase III Clinical Research, Fall River, Massachusetts
  - David S. Rosenberg, M.D, Florissant, Missouri
  - Dr Melvin Albert Churchill Jr, Lincoln, Nebraska
  - Prospect Medical Offices, Midland Park, New Jersey
  - Advanced Arthritis Care Center, Brooklyn, New York
  - Prem C.Chatpar, M.D., LLC, Plainview, New York
  - Box Arthritis and Rheumatology, Charlotte, North Carolina
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, North Charleston, South Carolina
  - Comprehensive Rheumatology Care, Hendersonville, Tennessee
  - Elizabeth Marini Simpson, Hixon, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Accurate Clinical Research, Houston, Texas
  - Clinical Research Institute of Houston, Houston, Texas
  - Spring Clinical Research, Tomball, Texas
  - Center for Arthritis and Rheumatic Diseases, P.C., Chesapeake, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (11):
  - Hospital Británico de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Sociedad Italiana de Beneficencia en Buenos Aires (Hospital Italiano de Buenos Aires), Ciudad Autónoma de Buenos Aires / Buenos Aires, Buenos Aires / Argentina
  - Instituto de Asistencia Reumatológica Integral I.A.R.I, San Fernando, Buenos Aires / Argentina
  - Clínica Adventista Belgrano, Ciudad Autónoma de Buenos Aires / Buenos Aires, Ciudad Autónoma de Buenos Aires / Buenos Aires /Argentina.
  - CIER, centro de investigaciones en enfermedades reumáticas (Razón social: ARIES MEDICA S.R.L.), Ciudad de Buenos Aires / Buenos Aires, Ciudad de Buenos Aires, Buenos Aires, Argentina
  - Sociedad Española de Beneficiencia y Mutualidad Hospital español de Mendoza, Godoy Cruz, Mendoza / Argentina
  - DIM Clinica Privada, Ramos Mejía, Ramos Mejía / Buenos Aires / Argentina
  - Centro Integral de Reumatología S.R.L., S.M. de Tucumán / Tucumán, S.M. de Tucumán / Tucumán / Argentina.
  - C.E.R - Centro Polivalente de Asistencia e Investigación Clínica propiedad de CER SAN JUAN S.R.L., San Juan, San Juan / San Juan / Buenos Aires
  - Instituto CAICI SRL., Rosario, Santa Fe / Argentina
  - I.N.Ne.L S.R.L. (Instituto de Neurología y Neurorrehabilitación del Litoral S.R.L.), Santa Fé, Santa Fé / Argentina
- Southern Clinical Research Pty Ltd, Sandy Bay, Hobart, Tasmania, Australia
- Bulgaria (4):
  - MHAT Burgas, Burgas
  - DCC Sveti Pantaleimon OOD, Pleven
  - MHAT Kaspela EOOD, Plovdiv
  - UMHAT "Sv.Ivan Rilski", Sofia
- Turkey (Türkiye) (4):
  - Cukurova Universitesi Tip Fakultesi Balcalı Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ataturk Universitesi Yakutiye Egitim ve Arastirma Hastanesi, Erzurum
  - Osmangazi Universitesi Tıp Fakultesi Hastanesi, Eskişehir

REFERENCES:
- [Derived] Bassiouni H, Spargo CE, Vlahos B, Jones HE, Pedersen R, Shirazy K. Maintenance of Remission with Etanercept-DMARD Combination Therapy Compared with DMARDs Alone in African and Middle Eastern Patients with Active Rheumatoid Arthritis. Rheumatol Ther. 2018 Jun;5(1):149-158. doi: 10.1007/s40744-018-0094-6. Epub 2018 Feb 26. PMID 29480357
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801364&StudyName=Drug%20Concentration%2C%20Immunogenicity%2C%20and%20Efficacy%20Study%20in%20Patients%20with%20Rheumatoid%20Arthritis%20Currently%20Treated%20with%20Etanercept%2C%20Adalimumab

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter, non-interventional (NI) study conducted to evaluate data collected from a cross sectional population of participants with rheumatoid arthritis (RA) who received treatment with etanercept, adalimumab, or infliximab for a minimum of 6 months and maximum of 24 months prior to the study assessment visit.
Pre-assignment Details: Participants treated with one of the three targeted therapies were enrolled using interactive response technology to assure data for approximately 200 participants were included for each RA treatment.
Groups:
- Etanercept: Participants who had received treatment with etanercept for a minimum of 6 months and maximum of 24 months prior to the study assessment visit.
- Adalimumab: Participants who had received treatment with Adalimumab for a minimum of 6 months and maximum of 24 months prior to the study assessment visit.
- Infliximab: Participants who had received treatment with infliximab for a minimum of 6 months and maximum of 24 months prior to the study assessment visit.
Period: Overall Study
Arm/Group | Etanercept | Adalimumab | Infliximab
Started | 202 | 199 | 204
Completed | 200 | 199 | 196
Not Completed | 2 | 0 | 8
Not completed — Incorrect diagnosis of RA | 0 | 0 | 1
Not completed — Received treatment for < 6 months | 0 | 0 | 1
Not completed — Received treatment for >24 months | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) composed of participants who had diagnosis of RA and who received treatment with etanercept, adalimumab, or infliximab for a minimum of 6 months and a maximum of 24 months prior to the study visit. Data was not collected or analyzed on participants who entered the study but did not complete based on not meeting criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Adalimumab | Infliximab | Total
Number analyzed (Participants) | 200 | 199 | 196 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.37) | 54.3 (12.95) | 60.7 (13.01) | 57.1 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 162 | 157 | 474
  Male | 45 | 37 | 39 | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Positive for Antidrug Antibodies Among Those Treated With Etanercept Versus Those Treated With Monoclonal Antibodies (Adalimumab or Infliximab).
Description: Percentage of participants positive for antidrug antibodies among those treated with etanercept versus those treated with monoclonal antibodies (adalimumab or infliximab) was determined.
Time Frame: 1 day
Population: FAS included participants who were diagnosed of RA and who received continuous treatment with either etanercept, adalimumab, or infliximab for a minimum of 6 months to 24 months prior to study assessment visit.
Measure: Number; unit: Percentage of participants
Groups:
- Adalimumab/ Infliximab: Participants who had received treatment with adalimumab or infliximab for a minimum of 6 months and maximum of 24 months prior to the study assessment visit.
Arm/Group | Etanercept | Adalimumab/ Infliximab
Number analyzed (Participants) | 200 | 394
Percentage of participants | 0 | 24.4
Statistical Analysis 1: Comparison: Etanercept vs Adalimumab/ Infliximab; This sample was to provide >95% power to detect a difference of 12% in the proportion of participants positive for antidrug antibodies between the group of participants treated with a soluble receptor TNF inhibitor (etanercept) and the group of participants treated with mAB TNF inhibitors (adalimumab and infliximab) (5% vs 17%, respectively), using a Chi square test with continuity correction, an alpha of 0.05, and attrition rate of 15%; Test type: Superiority or Other; p < 0.0001, Fisher Exact — As there was only one primary endpoint, no adjustment was made for multiple comparisons; Logistic regression was to be used but the model was not fit as there were no antibodies in the etanercept group. Fisher's exact test was used

2. Secondary Outcome: Percentage of Participants With Low Disease Activity (LDA) (DAS28 ESR Score ≤ 3.2) Among Those Who Are Antidrug Antibody Positive Versus Negative (All Patients Receiving Etanercept, Adalimumab, or Infliximab Combined).
Description: Percentage of participants with Low Disease Activity (LDA) (Disease Activity Score based on a 28-joint count [DAS28] Erythrocyte sedimentation rate [ESR] score ≤3.2) among those who are antidrug antibody positive versus negative (all participants receiving etanercept, adalimumab, or infliximab combined).
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- % AA+: Proportion of participants positive for antidrug antibodies among those treated with etanercept versus those treated with monoclonal antibodies (adalimumab or infliximab)
- % AA-: Proportion of participants negative for antidrug antibodies among those treated with etanercept versus those treated with monoclonal antibodies (adalimumab or infliximab)
Arm/Group | % AA+ | % AA-
Number analyzed (Participants) | 94 | 484
percentage of participants | 56.4 | 62.0

3. Secondary Outcome: Serum Trough Drug Concentrations for Etanercept, Adalimumab, and Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: Serum trough drug concentrations for etanercept, adalimumab, and infliximab compared between participants who are antidrug antibody positive versus negative. Units of measurement for Serum trough drug concentration is µg/mL.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 195
µg/mL
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 1.5 (2.24) | 0.2 (0.90)
  AA- | 1.8 (1.03) | 7.7 (4.72) | 9.8 (15.25)

4. Secondary Outcome: Percentage of Participants Positive for Antidrug Antibodies Among Those Treated With Etanercept, Adalimumab, or Infliximab.
Description: Percentage of participants positive for antidrug antibodies among those treated with etanercept, adalimumab, or infliximab were determined.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 195
Percentage of participants | 0 | 31.2 | 17.4

5. Secondary Outcome: The Clinical Disease Activity Index (CDAI) Total Scores for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: The CDAI total scores for etanercept, adalimumab, or infliximab compared between participants who are antidrug antibody positive versus negative. CDAI = Disease activity score (DAS) 28 prorated Swollen Joint Count (0-28) + DAS 28 prorated Tender Joint Count (0-28) + Physician's Global Assessment (0-10) + Subject's Global Assessment (0-10). The total score range is 0-76. Score interpretation: Remission ≤ 2.8; Low Disease Activity CDAI > 2.8 and ≤ 10; Moderate Disease Activity CDAI > 10 and ≤ 22; High Disease Activity CDAI > 22.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 194
units on a scale
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 17.3 (13.56) | 21.7 (16.12)
  AA- | 12.6 (10.62) | 16.3 (14.83) | 18.5 (13.84)

6. Secondary Outcome: The Simplified Disease Activity Index (SDAI) Total Scores for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: The SDAI Total Scores for etanercept, adalimumab, or infliximab compared between participants who are antidrug antibody positive versus negative. SDAI = DAS 28 prorated Swollen Joint Count (0-28) + DAS 28 prorated Tender Joint Count (0-28) + Physician's Global Assessment (0-10) + Subject's Global Assessment (0-10) + C-reactive protein (CRP) (in mg/dL). The total score range is 0-86. Score interpretation: Remission SDAI ≤ 3.3; Low Disease Activity SDAI > 3.3 and ≤ 11; Moderate Disease Activity SDAI > 11 and ≤ 26; High Disease Activity SDAI > 26.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 193
units on a scale
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 18.5 (14.52) | 23.1 (16.33)
  AA- | 13.5 (10.95) | 16.8 (14.91) | 19.2 (13.89)

7. Secondary Outcome: Disease Activity Score Based on a 28-joint Count (DAS28), Calculated With Erythrocyte Sedimentation Rate for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: The DAS28 assessment is a derived measurement with differential weight given to each component. DAS28 will be calculated twice, utilizing first ESR, and then CRP as the acute phase reactant: 1) DAS28-ESR = 0.56 sqrt (28 painful/tender joint count) + 0.28 sqrt (28 swollen joint count) + 0.70 (ln ESR) + 0.014 GH, where GH=subject general health VAS (0-100 mm). 2) DAS28-4 CRP = 0.56 sqrt (28 painful/tender joint count) + 0.28 sqrt (28 swollen count) + 0.36 (ln CRP+1) + 0.014 GH + 0.96, where GH=subject general health VAS (0- 100 mm), higher scores were indicative of a worse outcome. The specific components of the DAS28 assessment that were used in this study are: Tender/Painful Joint Count (28), Swollen Joint Count (28), ESR/CRP, and Subject's General Health VAS assessment.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 197 | 197 | 185
Units on a scale
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 3.1 (1.22) | 3.5 (1.33)
  AA- | 2.5 (1.20) | 2.8 (1.43) | 3.1 (1.31)

8. Secondary Outcome: Disease Activity Score, 28 Joint Count, Calculated With C-reactive Protein (DAS28-CRP) for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: The DAS28 assessment is a derived measurement with differential weight given to each component. DAS28 will be calculated twice, utilizing first ESR, and then CRP as the acute phase reactant: 1) DAS28-ESR = 0.56 sqrt (28 painful/tender joint count) + 0.28 sqrt (28 swollen joint count) + 0.70 (ln ESR) + 0.014 GH, where GH=subject general health VAS (0 100 mm). 2) DAS28-4 CRP = 0.56 sqrt (28 painful/tender joint count) + 0.28 sqrt (28 swollen count) + 0.36 (ln CRP+1) + 0.014 GH + 0.96, where GH=subject general health VAS (0-100 mm), higher scores were indicative of a worse outcome. The specific components of the DAS28 assessment that were used in this study are: Tender/Painful Joint Count (28), Swollen Joint Count (28), ESR/CRP, and Subject's General Health VAS assessment.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 195
Units on a scale
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 3.4 (1.22) | 3.7 (1.30)
  AA- | 2.9 (1.18) | 3.1 (1.36) | 3.4 (1.26)

9. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ DI) Scores for for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: The HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question in the questionnaire, the level of difficulty is scored from 0 to 3 with 0 representing "no difficulty," 1 as "some difficulty," 2 as "much difficulty," and 3 as "unable to do." Any activity that requires assistance from another individual or requires the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. The total score range for the HAQ-DI scale, minimum score was 0 (best), maximum score was 3 (worst).
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 195
Units on a scale
  AA+ | NA (NA) — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 1.0 (0.75) | 1.2 (0.69)
  AA- | 0.8 (0.68) | 0.9 (0.70) | 1.0 (0.63)

10. Secondary Outcome: Percentage of HAQ DI (<=0.5) Scores for Etanercept, Adalimumab, or Infliximab Compared Between Participants Who Are Antidrug Antibody Positive Versus Negative.
Description: HAQ DI (<=0.5) scores for etanercept, adalimumab, or infliximab compared between participants who are antidrug antibody positive versus negative.
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 200 | 199 | 195
percentage of participants
  % AA+ | NA — There were no participants in ETN arm tested positive for anti-etanercept antibody. | 30.6 | 20.6
  % AA- | 42.5 | 36.5 | 26.1

11. Secondary Outcome: Correlation of Antidrug Antibody Titers With Efficacy Measures.
Description: Correlation of antidrug antibody titers with efficacy measures analysed using Spearman correlation coefficient.
Time Frame: 1 day
Population: FAS included participants who were diagnosed of RA and who received continuous treatment with either etanercept, adalimumab, or infliximab for a minimum of 6 months to 24 months prior to study assessment visit. No participants for etanercept arm were antibody positive, therefore there is no correlation to report.
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 0 | 199 | 195
Correlation coefficient
  CDAI |  | 0.07447 | 0.05256
  SDAI |  | 0.08970 | 0.06806
  DAS28-ESR |  | 0.12179 | 0.08950
  DAS28-CRP |  | 0.12710 | 0.08366

12. Secondary Outcome: Correlation of Antidrug Antibody Titers With Trough Drug Concentration.
Description: Correlation of antidrug antibody titers with trough drug concentration analysed using Spearman correlation coefficient.
Time Frame: 1 day
Population: as for outcome 11
Measure: Number; unit: Correlation coefficient
Arm/Group | Etanercept | Adalimumab | Infliximab
Number analyzed (Participants) | 0 | 199 | 195
Correlation coefficient |  | -0.69017 | -0.60542

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent until the follow-up visit (+28 days) following the assessment visit.
Arm/Group | Etanercept | Adalimumab | Infliximab
Serious Adverse Events (participants affected / at risk) | 1/200 | 0/199 | 1/196
Other Adverse Events (participants affected / at risk) | 5/200 | 4/199 | 11/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=200) | Adalimumab (N=199) | Infliximab (N=196)
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Blood Count Abnormal (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=200) | Adalimumab (N=199) | Infliximab (N=196)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 2 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.